CLINICAL TRIAL: NCT02618746
Title: Home Rehabilitation Via Telemonitoring of Vital Signs to Prevent Exacerbations in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Home Rehabilitation Via Telemonitoring in Patients With COPD
Acronym: TELECARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thorax Research Foundation (Other)
Collaborators: National and Kapodistrian University of Athens (Other); Greek Ministry of Development (Other Government)
Responsible Party: Principal Investigator, IOANNIS VOGIATZIS, Associate Professor, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11SYN_10_1438
Record Dates: First submitted 2015-11-28; First posted 2015-12-01 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Telemonitoring; Home Rehabilitation; Exacerbations; Physical Activity; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A, Telerehabilitation (Experimental): The 12-month home care/rehabilitative program will include the following components: a) individualized action plan; b) educational session on self management; c) physical exercise sessions to remote monitoring; d) access to the call centre; e) professional weekly calls by physiotherapists, dietician and physician with remote connection as a response to possible incidents; f) remote monitoring selectively and temporarily.
  Interventions: Other: Telerehabilitation
- Group B, Hospital based Rehabilitation (Active Comparator): Patients assigned to the hospital based program will visit the hospital twice weekly for 12 months in order to participate in a multidisciplinary rehabilitation program including exercise, physiotherapy dietary and psychological advice by the staff of the rehabilitation centre based at the University clinic.
  Interventions: Other: Hospital based Rehabilitation
- Group C, Usual care Group (No Intervention): The control group will follow the usual care not involving the initial 8-week rehabilitation program neither maintenance hospital rehabilitation sessions or home telemonitoring of vital signs.

INTERVENTIONS:
Other: Telerehabilitation
  Arms: Group A, Telerehabilitation
Other: Hospital based Rehabilitation
  Arms: Group B, Hospital based Rehabilitation

SUMMARY:
COPD is the fourth leading cause of death in the world and is the only one of the top five illnesses whose death rate is still increasing. It is mainly caused by smoking. Greece has a higher prevalence and death rate for COPD than many other countries in Europe. The disease is incurable so treatment is aimed at alleviating symptoms and slowing progression. Despite maximal medication and strategies such as pulmonary rehabilitation and home nurse support, many patients remain vulnerable, socially isolated and report difficulty in accessing their local health services. Research has shown that patients have worsening symptoms for an average of three to four days before they are admitted to hospital with an exacerbation of COPD. This suggests a window of opportunity to intervene. Early warning and contact via innovative technology may treat symptoms earlier, improve patient confidence / quality of life and simultaneously reduce health care visits or admissions. However, there is a large gap between the postulated and empirically demonstrated benefits of electronic Health Technologies. In addition, there is a lack of robust research on the risks of implementing these technologies and their cost-effectiveness has yet to be demonstrated, despite being frequently promoted by policymakers as if this was a given issue. In addition, the evidence-base for telehealth is not well-reported in peer reviewed journals and hence there continue to be difficulties experienced in convincing clinicians, hospital managers and stakeholders that investment in such technologies will enable reductions in other aspects of healthcare delivery over time.

This project attempts to provide robust justification of the effectiveness of telerehabilitation by the implementation of a randomized controlled trial blindly assigning COPD patients to: i) a home care and telerehabilitation group remotely monitored by a specialised private health care centre (Filoktitis - group A) or ii) a hospital-based rehabilitation group managed at a regular base through weekly visits by personnel at a state University rehabilitation centre (group B). iii) A third group that receives usual care (group C: control group; i.e.: neither home monitoring nor hospital based rehabilitation) is also included.

DETAILED DESCRIPTION:
COPD is an important health problem in Greece as the average prevalence of COPD in people > 35 years old is 8.4% (i.e.: approximately 350.000 citizens) (Tzanakis et al., 2004). Hospitalization attributed to severe exacerbations is the major cost driver of COPD. A study in Northern Greece revealed that mean actual cost per severe exacerbation of COPD is €1711, whilst only the amount of €621 is reimbursed by social security funds (Geitona et al., 2011). The observed price discrepancies between the actual and the nominal cost per patient, undoubtedly increases public debt especially when considering that patients with severe COPD suffer from acute exacerbations twice or three times per year.

Accordingly, there is urgent need to prevent exacerbations and subsequent hospitalizations in Greece. International evidence supports the concept that telemonitoring has a key role to play in systemic improvements to healthcare by reducing unplanned hospital admissions, hospital length of stay and the use of health care services, thereby making best use of scarce clinical resources and empowering individual patients. Home telemonitoring of chronic lung diseases appears as a promising patient management approach that could potentially produce accurate and reliable data, empower patients, influence their attitudes and behaviour, and improve patients medical conditions.

However, the scientific evidence in support of home telemonitoring is still weak and inconsistent, which highlights the need for more research, particularly in relation to the patient-level benefits, associated with these technologies. Furthermore, although, economic viability of telemonitoring has been observed in very few studies, in most cases no in-depth cost-minimization analyses were performed (Casas et al., 2006; Hernandez et al., 2015). Accordingly, there is a need of studies to accumulate evidence related to the interaction between the clinical effects of telemonitoring, its cost effectiveness, the impact on services utilization, and acceptance by health care providers. The project looks into the sustainability of patient telemonitoring services implemented by a private health care enterprise, namely the Filoktitis Rehabilitation Centre and its clinical effectiveness compared to a long term program of hospital-based rehabilitation (at Athens University 1st Department of Respiratory Medicine) not requiring home telemonitoring. The proposed strategy will allow the analysis and evaluation of reimbursement schemes and the design of appropriate business models.

The main idea is to initially (8-weeks) teach COPD patients techniques of self-management and improve their functional capacity by regular exercise training taking place at two different rehabilitation centres (one state hospital: Athens University Clinic of Respiratory Medicine, and one private hospital: Filoktitis Rehabilitation Centre) and subsequently either have the patients visiting the State University Hospital twice weekly for wellness and rehabilitation sessions and for regular checking of their clinical condition for 12 months or in the case of Filoktitis refer patients home to live independently whilst remotely monitoring the course of a number of vital signs that alert the physician when an exacerbation is eminent. (i.e., prematurely recognize symptoms of exacerbation). The initial 8-week sessions of rehabilitation takes place at both the University Hospital Clinic and at Filoktitis rehabilitation centre, whilst home monitoring will be implemented only to those who complete the initial 8-week phase at Filoktitis Rehabilitation Centre for a subsequent period of 12 months. Patients who complete the initial 8-week program at the University Clinic will keep visiting the centre twice weekly for 12 months. The ultimate objective of this project is to identify, in terms of health status outcomes, patient compliance and cost effectiveness, whether remote monitoring and management of patients by professionals at the private rehabilitation centre is superior to that not involving telemonitoring but regular visits to the University Hospital Clinic.

The aim of the proposed project in terms of specific patient outcome measures (namely annual rate of hospital admissions due to an exacerbation and exacerbations treated at home, emergency room visits, use of health care resources, quality of life, functional capacity and daily levels of physical activity) to test the efficacy of wireless systems for patient's home self-monitoring when this service is delivered remotely by a private rehabilitation centre compared to close monitoring of patients through regular visits to the University Hospital Clinic.

The hypothesis to be tested will be that once the technology and knowledge is transferred to a private rehabilitation centre, patient follow-up and early prevention of exacerbations will not differ when patients are controlled remotely via home telemonitoring services compared to the management of patients at centralized Hospital level, since in the case of the latter type of service there are difficulties for elderly and frail patients to regularly visit the Hospital.

Study design: One hundred fifty (150) clinically stable patients classified by GOLD as stages II III and IV are recruited from the University Hospital Outpatient Clinic and the Filoktitis Medical Centre.

The study is conducted as a randomized controlled trial blindly assigned using a set of computer-generated random numbers to home care (group A, Telerehabilitation group: controlled by Filoktitis rehabilitation centre) or group B (Hospital based Rehabilitation supervised by the University hospital personnel) and a third group that will receive usual care (group C, usual care: control group). Prior to recruitment COPD patients initially complete a multidisciplinary intense Pulmonary Rehabilitation Program lasting for 8 weeks either at Filoktitis rehabilitation centre or at the University clinic rehabilitation centre at Sotiria Hospital (1st Department of Respiratory Medicine) to improve the functional capacity and quality of life. Thereafter patients assigned into group A (n = 50) are monitored at home for 12 months or for Group B (n= 50) followed by the University clinic professional twice weekly where visits to the hospital are scheduled for 12 months to undertake physiotherapy, dietary and psychological advice and exercise training sessions. The control group (C: = 50 patients) follows the usual care treatment not involving maintenance hospital rehabilitation sessions or home telemonitoring of vital signs.

The home care/rehabilitative program includes the following components: a) individualized action plan; b) educational session on self management; c) physical exercise sessions to remote monitoring; d) access to the call centre; e) professional monthly home visits of physiotherapists, dietician and physician with remote connection as a response to possible incidents; f) remote monitoring selectively and temporarily. The home care program will be performed by staff employed by Filoktitis rehabilitation centre.

Study protocol: On a daily basis, patients being recruited to the home care program (Telerehabilitation, group A) take one or more of their own vital sign measurements using wireless devices in their home. They may also manually enter some measurements into a tablet. Results are automatically transmitted from the tablet (via mobile communication network) to a secure web-based server platform, the in-home communication device that also prompts patients to answer clinician-directed health and risk assessment survey questions. A care management team based at Filoktitis (nurse or physician) reviews each patient's information on a web-based clinical review platform, and sends an alert to the patient's doctor when a vital sign measurement or survey response falls outside established limits. In addition to monitoring the tell-tale symptoms of decline - such as abnormal weight gain, increased blood pressure, shortness of breath, fatigue, or oedema, fever, cough - the system also triggers automated health assessments. Patients in group A are also given tasks to exercise regularly at home as well as they are remotely provided with dietary and psychological advice. Patients assigned to the hospital based rehabilitation program (group B) visit the hospital twice weekly for 12 months in order to participate to a multidisciplinary rehabilitation program including exercise, physiotherapy dietary and psychological advice by the staff of the rehabilitation centre based at the University clinic.

Outcomes assessed at 12 months follow up for all 3 groups: i) state of health evaluated with standardised questionnaires; ii) number of emergency room visits and unscheduled hospital admissions due to any cause; iii) annual rate of admitted days; iv) functional capacity); v) daily symptoms; vi) daily physical activity; vii) health-related quality of life. Frequency of assessment: outcomes will be assessed at baseline (prior to joining the initial 8 week rehabilitation program), at 6 months and 12 months following completion of the initial 8-weeks rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion in this study Patients fulfil all of the following criteria:

1. Written informed consent obtained before any assessment is performed.
2. Male and female patients ≥ 40 years of age
3. Diagnosis of COPD [post-bronchodilator forced expiratory volume at one second (FEV1) <80% predicted and FEV1/ forced vital capacity (FVC) <75% without significant post-bronchodilator reversibility (<10% FEV1 % predicted normal)]
4. Optimal medical treatment according to GOLD without regular use of systemic corticosteroids
5. Current or ex-smokers with a smoking history equivalent to at least 10 pack years (1 pack year = 20 cigarettes smoked per day for 1 year)
6. Absence of other significant diseases that could contribute to exercise limitation
7. At least 2 COPD exacerbations the year before the time entry

Exclusion Criteria:

Patients fulfilling any of the following criteria are not eligible for inclusion in this study. No additional exclusions are applied by the investigator, in order to ensure that the study population will be representative of all eligible patients.

1. Orthopedic, neurological or other complaints that significantly impair normal biomechanical movement patterns, as judged by the investigator. Specifically if the patients' condition/ co-morbidities are such that physical activity cannot be increased.
2. Respiratory diseases other than COPD (e.g. asthma)
3. Cognitive reading impairment and/or difficulties to manage electronic devices precluding interaction with the tablet, as judged by the investigator
4. Patients not on optimal pharmacotherapy
5. No COPD exacerbations the year before the time entry

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of exacerbations | 12 months
  Unscheduled hospital admissions due to an exacerbation including exacerbations treated at home

SECONDARY OUTCOMES:
Functional Capacity | 12 months
  6 min walk test
Number of visits to Emergency Outpatient Clinic | 12 months
Daily physical activity levels | 12 months
  Activity monitoring via accelerometers
Quality of life and symptoms | 12 months
  Questionaires

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Vogiatzis, Ph.D., Study Chair — National and Kapodistrian University of Athens

REFERENCES:
- [Background] Casas A, Troosters T, Garcia-Aymerich J, Roca J, Hernandez C, Alonso A, del Pozo F, de Toledo P, Anto JM, Rodriguez-Roisin R, Decramer M; members of the CHRONIC Project. Integrated care prevents hospitalisations for exacerbations in COPD patients. Eur Respir J. 2006 Jul;28(1):123-30. doi: 10.1183/09031936.06.00063205. Epub 2006 Apr 12. PMID 16611656
- [Background] Tzanakis N, Anagnostopoulou U, Filaditaki V, Christaki P, Siafakas N; COPD group of the Hellenic Thoracic Society. Prevalence of COPD in Greece. Chest. 2004 Mar;125(3):892-900. doi: 10.1378/chest.125.3.892. PMID 15006947
- [Background] Geitona M, Hatzikou M, Steiropoulos P, Alexopoulos EC, Bouros D. The cost of COPD exacerbations: a university hospital--based study in Greece. Respir Med. 2011 Mar;105(3):402-9. doi: 10.1016/j.rmed.2010.09.020. PMID 20970310
- [Background] Hernandez C, Alonso A, Garcia-Aymerich J, Grimsmo A, Vontetsianos T, Garcia Cuyas F, Altes AG, Vogiatzis I, Garasen H, Pellise L, Wienhofen L, Cano I, Meya M, Moharra M, Martinez JI, Escarrabill J, Roca J. Integrated care services: lessons learned from the deployment of the NEXES project. Int J Integr Care. 2015 Mar 30;15:e006. doi: 10.5334/ijic.2018. eCollection 2015 Jan-Mar. PMID 26034465
- [Derived] Poot CC, Meijer E, Kruis AL, Smidt N, Chavannes NH, Honkoop PJ. Integrated disease management interventions for patients with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2021 Sep 8;9(9):CD009437. doi: 10.1002/14651858.CD009437.pub3. PMID 34495549
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633
- [Derived] Vasilopoulou M, Papaioannou AI, Kaltsakas G, Louvaris Z, Chynkiamis N, Spetsioti S, Kortianou E, Genimata SA, Palamidas A, Kostikas K, Koulouris NG, Vogiatzis I. Home-based maintenance tele-rehabilitation reduces the risk for acute exacerbations of COPD, hospitalisations and emergency department visits. Eur Respir J. 2017 May 25;49(5):1602129. doi: 10.1183/13993003.02129-2016. Print 2017 May. PMID 28546268